CLINICAL TRIAL: NCT01300936
Title: Abdominal Wall Hernias and Abdominal Wall Function: A Quantitative Study of Trunk Strength.
Brief Title: Trunk Strength Study
Status: Completed | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: John Scott Roth, MD, University of Kentucky Medical Center
Other Study IDs: 09-0876-P6H
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Ventral/Incisional Hernia Repairs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with abdominal wall hernias

SUMMARY:
The purpose of this study is to measure abdominal wall strength both preoperatively and postoperatively in patients undergoing ventral/incisional hernia repairs. The investigators hypothesize that abdominal wall strength is improved in hernia repairs that reapproximate the rectus musculature to the midline. Abdominal wall strength measurements would be obtained utilizing various abdominal strength testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for hernia repair.

Exclusion Criteria:

* Pregnant females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo laparoscopic ventral hernia repair or open repair. People between the ages of 18 to 65 in relative good health.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-03

CONTACTS AND LOCATIONS:
Overall Officials: Scott Roth, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States